CLINICAL TRIAL: NCT03855878
Title: Prospective Observation of the Incidence and Natural History of Monoclonal Gammopathy in Patients Undergoing Weight Reduction Surgery
Brief Title: Observation of the Incidence and Natural History of MGUS in Patients Undergoing Weight Reduction Surgery
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rafat Abonour, Professor of Medicine, Indiana University
Other Study IDs: IUSCC-0633
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-10

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If patients are qualified for the study and elect to submit a sample for DNA it will be collected and stored at the Indiana biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Screening study to determine incidence of MGUS in this patient population

DETAILED DESCRIPTION:
This study is designed to observe the incidence of monoclonal gammopathy of undetermined significance (MGUS) among obese patients planning to have weight reduction surgery or planning to enter into a physician monitored weight loss program and to follow the regression or progression of MGUS following surgery or the initiation of the weight loss program.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 30 years or older planning to undergo weight reduction surgery or planning to enter into a physician monitored weight loss program
2. Patients must be obese, defined as a BMI ≥ 30 as calculated by the formula:

   weight in pounds / height squared x 703 = BMI
3. Subject consent and authorization for the release of health information must be obtained according to local institutional guidelines.
4. To remain in the study for the follow-up phase, the baseline screening test must indicate that a patient has MGUS.

Exclusion Criteria:

1. No history of any malignancy except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years.
2. No concurrent or planned participation in randomized trials of weight loss.
3. A patient will be excluded from the follow-up phase if the baseline screening test indicates they do not have MGUS

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To evaluate the incidence of MGUS in obese subjects 30 years and older planning to undergo weight reduction surgery or who have agreed to enter into a physician monitored weight loss program.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Rate of MGUS | 5 years
  The primary analysis focuses on the estimation of the rate of MGUS for this specific population.

CONTACTS AND LOCATIONS:
Overall Officials: Rafat Abonour, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared